CLINICAL TRIAL: NCT00697372
Title: SEA-SIDE: Sirolimus Versus Everolimus-eluting Stent Randomized Assessment in Bifurcated Lesions and Clinical SIgnificance of Residual siDE-branch Stenosis
Acronym: SEA-SIDE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Francesco Burzotta MD PhD, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P648
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Coronary Artery Disease; Coronary Stenosis
Keywords: Angioplasty, Transluminal, Percutaneous Coronary; Drug-Eluting Stents
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SES (Active Comparator): Patients with coronary bifurcation lesions treated by Sirolimus eluting stent
  Interventions: Device: Sirolimus eluting stent
- EES (Active Comparator): Patients with coronary bifurcation lesions treated by Everolimus eluting stent
  Interventions: Device: Everolimus eluting stent

INTERVENTIONS:
Device: Sirolimus eluting stent — Implantation of Sirolimus eluting stent
  Other Names: Cypher stent - Cordis (Johnson&Johnson Company)
  Arms: SES
Device: Everolimus eluting stent — Implantation of Everolimus eluting stent
  Other Names: Xience stent - Abbot company
  Arms: EES

SUMMARY:
BACKGROUND:

Bifurcated lesions are a challenging subset in percutaneous coronary interventions (PCI). The selection of the type of DES and the technique for stent implantation have not been clarified. The side-branch (SB) is emerging as critical point, accounting for more than a third of the significant restenosis in the DES era. A series of data supports the adoption of a conservative strategy: stenting the main vessel (MV) only and reserving a conservative approach on the SB. Yet, the clinical relevance in terms of inducible ischemia of sub-optimal angiographic result has not been clarified.

AIMS OF THE STUDY:

The aims of the present study are:

1. to compare in a prospective randomized study the acute 3D angiographic results and the late clinical outcome of Sirolimus-eluting (SES) vs Everolimus-eluting stent (EES) obtained using a provisional TAP-stenting technique.
2. to prospectively assess the clinical relevance (inducible ischemia) of suboptimal angiographic result in the SB after stenting.

METHODS TO BE APPLIED:

150 consecutive patients with bifurcated lesions undergoing PCI with the provisional TAP-stenting technique will be randomized to SES or EES implantation. Procedural and post-PCI details will be prospectively recorded. The subgroup of patients in which complete revascularization has been achieved will enter a systematic assessment of inducible ischemia by early and late exercise tests.

Off line 3D QCA assessment will be performed and used to divide the study population in 2 groups according to the SB residual stenosis:

* Group O (optimal SB angiographic result): post-PCI SB area stenosis<50%
* Group S (sub-optimal SB angiographic result): post-PCI SB area stenosis>50%.

PRIMARY STUDY END-POINTS.

1. COMPARISON BETWEEN SES AND EES:

   SB acute angiographic result; SB trouble; target bifurcation failure.
2. SB-RELATED ISCHAEMIA of Group O vs Group S in patients with complete revascularization: inducible ischemia at the early exercise test or occurrence of early spontaneous ischemia related to the SB.

DETAILED DESCRIPTION:
Bifurcated lesions are challenging target lesions in percutaneous coronary interventions (PCI) which may specifically benefit from the usage of drug-eluting stents (DES). However, the selection of the type of DES and the technique for DES implantation have not been clarified. In spite of the technique adopted, the side-branch (SB) is emerging as critical point, accounting for more than a third of the significant restenosis in the DES era. A series of data supports the adoption of a conservative strategy: stenting the main vessel (MV) only and reserving a conservative approach on the SB as this is not associated with worse outcome compared to more complex stenting strategies. Yet, the clinical relevance in terms of inducible ischemia of sub-optimal angiographic result has not been clarified.

AIMS OF THE STUDY:

The aims of the present study are:

1. to compare in a prospective randomized study the acute 3D angiographic results (as a measure of the impact of stent design) and the late clinical outcome of Sirolimus-eluting (SES) vs Everolimus-eluting stent (EES) obtained using a provisional TAP-stenting approach to treat bifurcated lesions.
2. to prospectively assess the clinical relevance (in terms of inducible ischemia) of suboptimal angiographic result in the SB of bifurcated lesions treated by stenting.

METHODS TO BE APPLIED:

150 consecutive patients with bifurcated lesions undergoing PCI with the provisional TAP-stenting technique will be randomized to SES or EES implantation. Procedural details, post-PCI cardiac enzyme release, clinical outcome up to 1 year will be prospectively recorded. After the procedure, the subgroup of patients in which complete revascularization has been achieved (no untreated stenosis >50% in any other vessel, no residual stenosis >50% in any other treated vessel), will enter a systematic assessment of inducible ischemia by early (<8 days) and late (6-month) exercise tests.

Off line 3D QCA assessment will be performed and used to divide the study population in 2 groups according to the SB residual stenosis: Group O (optimal SB angiographic result): post-PCI SB area stenosis<50% and Group S (sub-optimal SB angiographic result): post-PCI SB area stenosis>50%.

PRIMARY STUDY END-POINTS.

1. COMPARISON BETWEEN SES AND EES:

   * "SB acute angiographic result": comparison of the 3DQCA-estimated MLD and MLA in the SB.
   * "SB trouble": composite of: 1. occurrence of SB TIMI flow <3 after MV stenting throughout the procedure; 2. need of guidewire(s) different from BMW to re-wire SB after MV stenting; 3. failure to re-wire the SB after MV stenting; 4. failure to dilate the SB after MV stenting and SB re-wiring.
   * target bifurcation failure (TBF) defined as target bifurcation-related major adverse coronary events (MACE) or target bifurcation angiographic failure.
2. SB-RELATED ISCHAEMIA of Group O vs Group S in patients with complete revascularization: inducible ischemia (diagnostic ST-segment changes) at the early (<8 days) exercise test or occurrence of early (<12 weeks) spontaneous ischemia related to the SB (any ischemic episode requiring unplanned coronary angiography with documentation of main vessel patency).

ELIGIBILITY:
Inclusion Criteria:

* de novo bifurcated lesions
* lesions >50% located in a major bifurcation point
* TIMI >2 on both main vessel and side branch
* main vessel visual diameter >2.5 mm
* side branch visual diameter >2.0 mm
* >18 years of age
* signed the informed consent to enter the study

Exclusion Criteria:

* known hypersensitivity to Sirolimus, Everolimus, cobalt, chromium, nickel, tungsten acrylic and fluoro-polymers
* contraindications to double antiplatelet therapy acute (within 48 hours) ST-elevation acute myocardial infarction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-09; Primary Completion 2008-10 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
6-9-12-18 MONTH CLINICAL OUTCOME (Comparison of the rate of target bifurcation failure) | 18 MONTHS
ACUTE ANGIOGRAPHIC RESULT | 7 DAYS
  * "MV acute angiographic result": comparison of the 3DQCA-estimated MLD and MLA in the MV.
  * "SB acute angiographic result": comparison of the 3DQCA-estimated MLD and MLA in the SB.
SIDE BRANCH TROUBLE | 7 DAYS
  "SB trouble" composite of:
  1. occurrence of SB TIMI flow <3 after MV stenting throughout the procedure;
  2. need of guidewire(s) different from BMW to re-wire SB after MV stenting;
  3. failure to re-wire the SB after MV stenting;
  4. failure to dilate the SB after MV stenting and SB re-wiring.
TARGET BIFURCATION FAILURE | 18 MONTHS
  - target bifurcation failure (TBF) defined as target bifurcation-related major adverse coronary events (MACE) or target bifurcation angiographic failure.

SECONDARY OUTCOMES:
TECHNICAL CHARACTERISTICS | 7 DAYS
  comparison of procedural time, fluoroscopy time, total x-ray exposure, contrast media volume usage, number of guidewires used to wire the SB, direct stenting failure rate, kissing balloon rate, occurrence of transient deterioration of blood flow through the SB (TIMI<3)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Burzotta, MD,PhD,FESC, Principal Investigator — Catholic University of Sacred Heart
Locations (1):
- Institute of Cardiology - Catholic University of Sacred Heart, Rome, Italy

REFERENCES:
- [Background] Colombo A, Moses JW, Morice MC, Ludwig J, Holmes DR Jr, Spanos V, Louvard Y, Desmedt B, Di Mario C, Leon MB. Randomized study to evaluate sirolimus-eluting stents implanted at coronary bifurcation lesions. Circulation. 2004 Mar 16;109(10):1244-9. doi: 10.1161/01.CIR.0000118474.71662.E3. Epub 2004 Feb 23. PMID 14981005
- [Background] Ormiston JA, Webster MW, El Jack S, Ruygrok PN, Stewart JT, Scott D, Currie E, Panther MJ, Shaw B, O'Shaughnessy B. Drug-eluting stents for coronary bifurcations: bench testing of provisional side-branch strategies. Catheter Cardiovasc Interv. 2006 Jan;67(1):49-55. doi: 10.1002/ccd.20453. PMID 16003787
- [Background] Pan M, Suarez de Lezo J, Medina A, Romero M, Delgado A, Segura J, Ojeda S, Mazuelos F, Hernandez E, Melian F, Pavlovic D, Esteban F, Herrador J. Drug-eluting stents for the treatment of bifurcation lesions: a randomized comparison between paclitaxel and sirolimus stents. Am Heart J. 2007 Jan;153(1):15.e1-7. doi: 10.1016/j.ahj.2006.10.017. PMID 17174630
- [Background] Lefevre T, Louvard Y, Morice MC, Loubeyre C, Piechaud JF, Dumas P. Stenting of bifurcation lesions: a rational approach. J Interv Cardiol. 2001 Dec;14(6):573-85. doi: 10.1111/j.1540-8183.2001.tb00375.x. PMID 12053378
- [Background] Ge L, Tsagalou E, Iakovou I, Sangiorgi GM, Corvaja N, Airoldi F, Chieffo A, Montorfano M, Michev I, Colombo A. In-hospital and nine-month outcome of treatment of coronary bifurcational lesions with sirolimus-eluting stent. Am J Cardiol. 2005 Mar 15;95(6):757-60. doi: 10.1016/j.amjcard.2004.11.030. PMID 15757605
- [Background] Valgimigli M, Malagutti P, Rodriguez Granillo GA, Tsuchida K, Garcia-Garcia HM, van Mieghem CA, Van der Giessen WJ, De Feyter P, de Jaegere P, Van Domburg RT, Serruys PW. Single-vessel versus bifurcation stenting for the treatment of distal left main coronary artery disease in the drug-eluting stenting era. Clinical and angiographic insights into the Rapamycin-Eluting Stent Evaluated at Rotterdam Cardiology Hospital (RESEARCH) and Taxus-Stent Evaluated at Rotterdam Cardiology Hospital (T-SEARCH) registries. Am Heart J. 2006 Nov;152(5):896-902. doi: 10.1016/j.ahj.2006.03.029. PMID 17070153
- [Background] Iakovou I, Ge L, Colombo A. Contemporary stent treatment of coronary bifurcations. J Am Coll Cardiol. 2005 Oct 18;46(8):1446-55. doi: 10.1016/j.jacc.2005.05.080. Epub 2005 Sep 28. PMID 16226167
- [Background] Pan M, de Lezo JS, Medina A, Romero M, Segura J, Pavlovic D, Delgado A, Ojeda S, Melian F, Herrador J, Urena I, Burgos L. Rapamycin-eluting stents for the treatment of bifurcated coronary lesions: a randomized comparison of a simple versus complex strategy. Am Heart J. 2004 Nov;148(5):857-64. doi: 10.1016/j.ahj.2004.05.029. PMID 15523318
- [Background] Ge L, Iakovou I, Cosgrave J, Agostoni P, Airoldi F, Sangiorgi GM, Michev I, Chieffo A, Montorfano M, Carlino M, Corvaja N, Colombo A. Treatment of bifurcation lesions with two stents: one year angiographic and clinical follow up of crush versus T stenting. Heart. 2006 Mar;92(3):371-6. doi: 10.1136/hrt.2005.061531. Epub 2005 Jun 17. PMID 15964941
- [Background] Steigen TK, Maeng M, Wiseth R, Erglis A, Kumsars I, Narbute I, Gunnes P, Mannsverk J, Meyerdierks O, Rotevatn S, Niemela M, Kervinen K, Jensen JS, Galloe A, Nikus K, Vikman S, Ravkilde J, James S, Aaroe J, Ylitalo A, Helqvist S, Sjogren I, Thayssen P, Virtanen K, Puhakka M, Airaksinen J, Lassen JF, Thuesen L; Nordic PCI Study Group. Randomized study on simple versus complex stenting of coronary artery bifurcation lesions: the Nordic bifurcation study. Circulation. 2006 Oct 31;114(18):1955-61. doi: 10.1161/CIRCULATIONAHA.106.664920. Epub 2006 Oct 23. PMID 17060387
- [Background] Koo BK, Kang HJ, Youn TJ, Chae IH, Choi DJ, Kim HS, Sohn DW, Oh BH, Lee MM, Park YB, Choi YS, Tahk SJ. Physiologic assessment of jailed side branch lesions using fractional flow reserve. J Am Coll Cardiol. 2005 Aug 16;46(4):633-7. doi: 10.1016/j.jacc.2005.04.054. PMID 16098427
- [Background] Burzotta F, Gwon HC, Hahn JY, Romagnoli E, Choi JH, Trani C, Colombo A. Modified T-stenting with intentional protrusion of the side-branch stent within the main vessel stent to ensure ostial coverage and facilitate final kissing balloon: the T-stenting and small protrusion technique (TAP-stenting). Report of bench testing and first clinical Italian-Korean two-centre experience. Catheter Cardiovasc Interv. 2007 Jul 1;70(1):75-82. doi: 10.1002/ccd.21194. PMID 17585382
- [Background] Gradaus R, Mathies K, Breithardt G, Bocker D. Clinical assessment of a new real time 3D quantitative coronary angiography system: evaluation in stented vessel segments. Catheter Cardiovasc Interv. 2006 Jul;68(1):44-9. doi: 10.1002/ccd.20775. PMID 16770813
- [Derived] Burzotta F, Trani C, Todaro D, Lanza GA, Mariani L, Tommasino A, Niccoli G, Porto I, Leone AM, Crea F. Prospective evaluation of myocardial ischemia related to post-procedural side-branch stenosis in bifurcated lesions treated by provisional approach with drug-eluting stents. Catheter Cardiovasc Interv. 2012 Feb 15;79(3):351-9. doi: 10.1002/ccd.23218. Epub 2011 Dec 12. PMID 21735527
- [Derived] Burzotta F, Trani C, Todaro D, Mariani L, Talarico GP, Tommasino A, Giammarinaro M, Niccoli G, Porto I, Leone AM, Mongiardo R, Mazzari MA, Schiavoni G, Crea F. Prospective randomized comparison of sirolimus- or everolimus-eluting stent to treat bifurcated lesions by provisional approach. JACC Cardiovasc Interv. 2011 Mar;4(3):327-35. doi: 10.1016/j.jcin.2010.12.005. PMID 21435612
- [Derived] Sgueglia GA, Burzotta F, Trani C, Todaro D, Talarico GP, Niccoli G, Porto I, Leone AM, Coluccia V, Mazzari MA, Mongiardo R, Schiavoni G, Crea F. Comparative assessment of mammalian target of rapamycin inhibitor-eluting stents in the treatment of coronary artery bifurcation lesions: the CASTOR-Bifurcation registry. Catheter Cardiovasc Interv. 2011 Mar 1;77(4):503-9. doi: 10.1002/ccd.22714. PMID 20602477